CLINICAL TRIAL: NCT06989788
Title: A Randomised, Double-blind, Placebo-controlled, Single Centre, Phase I Study to Evaluate the Safety, Reactogenicity and Immunogenicity of AstriVax' Investigational Therapeutic Hepatitis B Virus (HBV) Vaccine (AVX70371) in Healthy Adults Aged 18 to 40 Years
Brief Title: A Study to Evaluate the Safety and Immunogenicity of an Investigational Vaccine for Chronic Hepatitis B Virus Infection, in Healthy Adults
Acronym: RUBY
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstriVax Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVX37-102; 2025-521169-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVX70371 (Experimental): Participants in this arm receive administrations of AVX70371
  Interventions: Biological: AVX70371
- Placebo (Placebo Comparator): Participants in this arm receive administrations of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AVX70371 — AstriVax Therapeutics' HBV immunotherapeutic
  Arms: AVX70371
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this first time in humans trial is to evaluate the safety, reactogenicity and immunogenicity of repeated administrations of AVX70371 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female assigned at birth, inclusive of all gender identities
* Between, and including, 18 and 40 years of age on the day of the Screening Visit
* Healthy individual, as established by the Investigator
* Able to read and understand the informed consent form, and written informed consent obtained from the participant
* Participants who, in the opinion of the Investigator, can and will comply with the requirements of the protocol

Exclusion Criteria:

* Body Mass Index < 18.0 or > 32.0 kg/m2
* Use of any investigational or non-registered product other than the study vaccination within 1 month preceding study entry, or concurrent participation in another clinical study in which the participant has been or will be exposed to an investigational or non-registered product, at any time during the study period
* Administration / planned administration of any vaccine not foreseen by the study protocol within 1 month preceding the first study vaccination and up to 1 month after the last study vaccination
* Presence of serologic marker of acute, chronic or past HBV infection
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months preceding first study vaccination, or planned chronic administration at any time during the study period
* Administration of long-acting immune-modifying drugs within 6 months or 5 half-lives (whichever is longer) preceding first study vaccination, or planned administration at any time during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history, family history or physical examination
* Administration of immunoglobulins and / or any blood or blood-derived products within 3 months preceding the first study vaccination, or planned administration during the study period
* History of or current autoimmune disease
* Malignancies or lymphoproliferative disorders within previous 5 years
* Personal or family history of thymic pathology
* History of any neurological disorders or seizures
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the investigational vaccine
* Moderate or severe acute disease in the opinion of the Investigator, and / or fever, on Day 1
* Alcohol, prescription drug, or substance (ab)use that, in the opinion of the Investigator, might interfere with the study conduct and / or participant safety
* Pregnant or lactating woman
* Woman of childbearing potential who is not utilizing a highly effective birth control method for at least 1 month prior to the first study vaccination, or who is planning to discontinue highly effective contraception prior to 2 months following the last study vaccination
* Employed by the Sponsor, by the contract research organisations working on behalf of the Sponsor, by the Investigator or the study site, or close relatives of research staff working on this study
* Medical condition or use of medication(s) that can increase the risk of bleeding or haematoma
* Any other condition or finding that the Investigator judges may interfere with study procedures or study results, or renders the participant unsuitable for the study

Note: other protocol-defined inclusion / exclusion criteria may apply.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited adverse events | During a 14-day follow-up period after each administration
Occurrence of unsolicited adverse events | From Day 1 up to 1 month after the last administration
Occurrence of hematological and biochemical laboratory abnormalities | From Day 1 up to 1 month after the last administration
Occurrence of adverse events of special interest | From Day 1 up to 1 year after the last administration
Occurrence of serious adverse events | From Day 1 up to 1 year after the last administration

SECONDARY OUTCOMES:
Cellular immune response following administrations of AVX70371, as measured by Intracellular Cytokine Staining (ICS) | From Day 1 up to 1 year after the last administration
Humoral immune response following administrations of AVX70371, as measured by enzyme-linked immunosorbent assay (ELISA) | From Day 1 up to 1 year after the last administration

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent - Centrum voor Vaccinologie (CEVAC), Ghent, Belgium